CLINICAL TRIAL: NCT00428051
Title: Multinational Latin American Epidemiologic Surveillance For Invasive Pneumococcal Disease
Brief Title: Colombia Epidemiologic Surveillance Study
Acronym: LEAP II
Status: Terminated | Type: Observational
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0887X1-900; B1841004
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Pneumonia; Meningitis; Bacteremia; Sepsis
Keywords: Epidemiology; Surveillance; Streptococcal Pneumonia
MeSH Terms: conditions — Pneumonia; Meningitis; Bacteremia; Sepsis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebral Spinal Fluid Pleural Fluid S. pneumoniae isolates
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All eligible patients
  Interventions: Other: Surveillance

INTERVENTIONS:
Other: Surveillance — No study drug, only interventions are blood draws and Chest X-rays

SUMMARY:
The study will determine the reduction in invasive pneumococcal disease (IPD) after the introduction of a National Immunization Program with PCV-7 in Bogota. The original LEAP study determine incidence of IPD prior to introduction of PCV-7 in Brazil, Costa Rica and Colombia. LEAP II is the continuation of the study in Colombia only.

DETAILED DESCRIPTION:
The study was stopped based on a decision to include PCV 10 in the National Immunization Program in Colombia. The study was designed to measure the impact of PCV 7 and 13 and is no longer feasible.

ELIGIBILITY:
Inclusion Criteria:

* Children 28 days to 36 months of age
* Presenting to a participating facility with a measured temperature of 39 degrees C or higher within 24 hours prior to screening, or with clinical suspicion of pneumonia, meningitis, bacteremia, sepsis, or other invasive pneumococcal disease

Exclusion Criteria:

* Any patient hat based on the clinical impression of the treating physician should not participate in the study: examples such as those with suspected dengue or urinary tract infection

Ages: 28 Days to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Epidemiologic study that will include children 28 days to 36 months of age that meet entrance criteria
Sampling Method: Probability Sample
Enrollment: 32867 (Actual)
Dates: Start 2006-09; Primary Completion 2011-02 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Annual age specific incidence rate of invasive pneumococcal disease based on the number of identified cases from the study sites and the size of the population at risk for children 28 days to 36 months of age | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Pfizer Investigational Site, Goiânia, Goiás, Brazil
- Pfizer Investigational Site, Bogotá, Colombia
- Pfizer Investigational Site, Uruca, Provincia de San José, Costa Rica

REFERENCES:
- [Derived] Benavides JA, Ovalle OO, Salvador GR, Gray S, Isaacman D, Rodgers GL. Population-based surveillance for invasive pneumococcal disease and pneumonia in infants and young children in Bogota, Colombia. Vaccine. 2012 Aug 31;30(40):5886-92. doi: 10.1016/j.vaccine.2012.03.054. Epub 2012 Apr 4. PMID 22484295
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0887X1-900&StudyName=Colombia%20Epidemiologic%20Surveillance%20Study